CLINICAL TRIAL: NCT00929214
Title: Aggressive Local Therapy for Limited Bone-Only Metastasis to Improve Progression-Free Survival in Breast Cancer Patients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0319; NCI-2011-02165 (Registry Identifier: NCI CTRP- Clinical Trials Registry)
Record Dates: First submitted 2009-06-25; First posted 2009-06-26 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Metastasized; Limited bone-only metastasis; Local Therapy; Radiation; Radiation Therapy; RT; Surgery; Standard Therapy; Chemotherapy; Endocrine Therapy
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Standard of Care; Drug Therapy; Neoadjuvant Therapy; Hyperthermia, Induced; Radiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (1):
- Standard Therapy + Local Therapy (Experimental): Systemic Standard Therapy (chemotherapy and/or endocrine therapy) + Local Therapy (surgery and/or radiation)
  Interventions: Drug: Standard Therapy; Procedure: Local Therapy

INTERVENTIONS:
Drug: Standard Therapy — Chemotherapy and/or Endocrine Therapy:
  For 3 - 9 months, all patients will receive systemic chemotherapy agents appropriate for the tumor characteristics and patient's prior treatment history, and may also be placed on endocrine therapy as determined by the treating medical oncologist.
  Other Names: Chemotherapy; Endocrine Therapy; Systemic Chemotherapy
Procedure: Local Therapy — Surgery and/or Radiation Therapy
  With no more than 3 bone metastases, local treatments including high-dose radiation therapy and/or surgery will be given. Radiation therapy involves daily treatments during weekdays that may last 5 to 7 weeks in a row. Each daily treatment may last 30 - 40 minutes. Surgery, including recovery, may last 4 to 6 weeks.
  Other Names: Radiation Therapy; RT; XRT; Surgery

SUMMARY:
The goal of this clinical research study is to find out if adding local therapy (surgery and/or radiation) to standard therapy (chemotherapy or endocrine therapy) in the treatment of patients with metastatic breast cancer can help to control the disease for a longer period of time than standard therapy alone.

DETAILED DESCRIPTION:
Study Treatments:

Current standard of care for breast cancer patients whose disease has spread to the bones is to treat them with chemotherapy or endocrine therapy. However, using radiation and surgery as well may help to get rid of the cancer cells in the bone lesions.

All participants will receive separate consent documents to sign that will explain the routine surgery, radiation therapy, and chemotherapy.

Standard Therapy:

If the imaging scans show that you are not at increased risk for bone fracture, you will receive 3 to 9 months of systemic therapy that is most appropriate for you as decided by your doctor. You may also be placed on endocrine therapy as decided by your doctor. If you have received drugs in the past that could cause heart-related side effects and/or a history of heart disease, you may have heart function tests, if your cancer doctor decides it is needed.

Study Visits:

After you have received 3-9 months of standard therapy, you will receive an MRI scan, a PET/CT scan, an X-ray, and a whole-body bone scan to make sure you still have no more than 3 bone metastases. Blood (about 2 tablespoons) and urine tests will also be collected to make sure you have no more than 3 bone metastases.

Local Therapy:

If you still have no more than 3 bone metastases, local treatments including high-dose radiation therapy and/or surgery will be given. The most appropriate local therapy will be chosen by your treating radiation oncologist, surgeon, and medical oncologist.

For bones with fractures or at risk for fracture, a rod or other devices may be placed in the bone to fix the bone. Radiation therapy involves daily treatments during weekdays that may last 5 to 7 weeks in a row. Each daily treatment may last 30 - 40 minutes. For special cases, shorter courses of radiation therapy may be offered to treat the lesions in the spine. Radiation types, such as photon, electron, or proton will be selected by your doctor.

If you have a risk of bone fracture due to the cancer, you may be treated with surgery and/or radiation first, before starting standard therapy. Again, the most appropriate local therapy will be chosen by your treating radiation oncologist, surgeon, and medical oncologist.

After completing the local therapies, you will receive an MRI scan, a PET/CT scan, a X-ray, and a whole-body bone scan to make sure you still have no more than 3 bone metastases. Blood (about 2 tablespoons) and urine will also be collected to make sure you have no more than 3 bone metastases. Then, you will receive 3 to 9 months of systemic therapy that is most appropriate for you as decided by your doctor. You may also be placed on endocrine therapy as decided by your doctor.

Length of Study:

The standard systemic therapy treatments may last 3 to 9 months. The radiation therapy process may last 6 to 8 weeks. Surgery, including recovery, may last 4 to 6 weeks. You will be taken off study early if you are found to have more than 3 lesions, if the disease worsens, or if you have intolerable side effects.

Long-Term Follow-up:

After the local and standard therapies are finished, you will have a follow-up visit at 3 months and every 3 months for the 1st year after the therapies, and then every 6 months for the 2nd and 3rd year after the therapies. At each of these visits, the following tests will be performed:

* You will have periodic tests which may include an MRI scan, a PET/CT scan, an X-ray, and a whole-body bone scan to check on the status of the disease. Your doctor will decide which tests you will need. The tests will be done every 3 months for the first year and then every 6 months for the next 2 years.
* Blood (about 2 tablespoons) and urine will be collected to check on the status of the disease.
* You will complete QOL questionnaires.

After the completion of the 36 month visit, you are encouraged to follow-up at any time after the last visit up to 1 year. Your doctor may request that you have an MRI scan, a PET/CT scan, an X-ray, and/or a whole-body bone scan to check on the status of the disease.

This is an investigational study. The use of local treatments (surgery and radiation therapy) to treat metastatic lesions of the bone is investigational. The use of chemotherapy and endocrine therapy is standard of care for breast cancer patients with metastases.

Up to 75 evaluable patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Breast cancer with metastasis to skeletal sites only
2. 1 to 3 bone metastatic sites (metastatic lesions in the same bone that are within 3 cm of each other are considered as one site)
3. KPS greater than or equals to 70
4. Absolute neutrophil count of > 1500 per microliter and platelet count > 100,000 per microliter; AST and alkaline phosphatase < = 2.5 X normal limits, bilirubin < = 1.5 x normal limits, calculated creatinine clearance > 50 ml/min using Cockcroft-Gault formula: CrCl male = (140-age) x (wt. in kg)/(Serum Cr x 72); CrCl female = 0.85 x (CrCl male)
5. Patients may or may not have started bis-phosphonates.
6. Patients who have received prior chemotherapy for their original breast cancer treatment are still eligible.
7. Previous use of systemic therapy for bone metastasis is allowable as long as the systemic therapy use fits within the treatment plan as described in Proposed Treatment/Study Plan. (If the patient received less than 3 - 9 months of systemic therapy previously, the use of additional systemic therapy may be necessary to fit within the treatment plan)
8. Treating physician assesses tumor to be sufficiently distant from sensitive structures to be able to achieve greater than or equal to 66 Gy. (i.e., spinal cord tolerance respected in vertebral body metastasis.
9. Patients with immanent risk of fracture(s) may receive local therapy prior to systemic therapy. Otherwise systemic therapy should be given first as outlined in abstract treatment study plan sections 1 and 2.

Exclusion Criteria:

1. Distant metastasis to organs (local recurrence and regional lymph node recurrence are not considered as distant metastasis) other than bone
2. Prior radiation to site(s) of distant metastasis of bone
3. History of scleroderma and systemic lupus erythematosus which increases the risk of toxicity from radiation treatment
4. Second primary malignancy (skin cancer other than melanoma allowed) that is disease free for less than 3 years
5. Premenopausal and postmenopausal (amenorrheic for less than 12 months) women with either a positive or no pregnancy test (serum or urine) at baseline within 7 days study enrollment. Postmenopausal women who are amenorrheic for more than 12 months do not require pregnancy test.
6. Women with child-bearing potential not using a reliable an appropriate contraceptive method.
7. Patients with child-bearing potential will agree to use contraception while on study and for 30 days from the date of the last therapy on protocol.
8. If the patient requires surgery of the bone metastasis, clinically serious comorbidities that render patient not medically fit for surgery (e.g. congestive heart failure, symptomatic coronary artery disease, cardiac arrhythmias and chronic lung disease not well controlled with medication; myocardial infarction within 12 months of enrollment)
9. Central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant to preclude informed consent or interfere with complying with protocol treatments.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-06-24 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Progression-Free Survival (PFS) | Study assessment at 9 Months
  Progression-free survival defined as 1) development of distant soft tissue or visceral metastasis at any time, 2) progression of bone lesion(s) that received planned local therapy (as defined by the imaging response criteria described by Hamaoka et al., and 3) development of new bone lesions after patient receives planned local therapy. Development of additional bone metastasis prior to receiving planned local therapy not be considered as event if the total number of bone metastasis is 3 or less. An event has occurred if additional bone metastasis develops and total number of bone metastasis is 4 or more.

CONTACTS AND LOCATIONS:
Overall Officials: Eric A. Strom, MD, BS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org